CLINICAL TRIAL: NCT06722378
Title: Bedside Notes: A Multicenter Trial to Improve Family Clinical Note Access and Outcomes for Hospitalized Children
Brief Title: A Trial to Improve Family Clinical Note Access and Outcomes for Hospitalized Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Pediatric Research in Inpatient Settings (PRIS) Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-1396; 1R01HS030098-01 (AHRQ); Protocol Version 2/6/2025 (Other: UW Madison); A536771 (Other: UW Madison)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hospitalized Child; Pediatric Patient Safety; Medical Errors; Parental Engagement in Care; Inpatient Pediatric Care
Keywords: Family-Centered Care; Electronic Health Records (EHR); Safety Reporting; Parent Note Access; Quality Improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to notes on a tablet (Experimental): Participants will be provided a tablet and will be able to access their child's medical notes while in the hospital.
  Interventions: Other: Access to medical notes
- Care as usual (No Intervention): Participants will not have access to a table to view their child's medical notes while in the hospital.

INTERVENTIONS:
Other: Access to medical notes — Inpatient notes shared in real-time on a hospital-owned bedside tablet linked to their child's records.
  Arms: Access to notes on a tablet

SUMMARY:
This study will test if giving parents access to their child's medical notes on a bedside tablet:

* helps them get more involved in their care
* helps identify safety concerns

Parents of hospitalized children will be randomly assigned to either use the Bedside Notes tool or follow usual care.

To see if this approach improves care and safety, researchers will measure:

* note access
* parent-reported safety concerns
* overall experiences

DETAILED DESCRIPTION:
Hospitalized children face alarming rates of harm due to medical errors, yet parents often lack access to the clinical information necessary to partner effectively in their child's care. Although clinicians are required to share inpatient clinical notes detailing diagnoses and treatment plans, <10% of parents access these notes during hospitalization. To address this critical gap, we developed the Bedside Notes intervention, a multicomponent strategy to improve parent access to clinical notes during their child's hospitalization and engage them in safety efforts. The intervention includes: (1) real-time access to inpatient notes through their child's patient portal on a bedside tablet and (2) a notes orientation video. In a single-center study, this intervention was associated with a >10-fold increase in parent note access and enabled 20% of parents to identify potential safety concerns, with 60% of these concerns confirmed as safety issues.

This multisite randomized controlled trial (RCT) will evaluate the effectiveness of the Bedside Notes intervention in improving parent access to inpatient notes and enhancing safety reporting. Specific aims are to: (1) assess the impact of the intervention on parent note access, (2) evaluate its effect on parent-reported safety concerns and experiences, and (3) identify barriers and facilitators to implementation. Guided by the Systems Engineering Initiative for Patient Safety 2.0 framework, this hybrid type 1 RCT will enroll English- and Spanish-speaking parents of 600 children admitted to pediatric services at three hospitals. Parents will be randomized to either: (1) usual care (access to outpatient portals on personal devices) or (2) the Bedside Notes intervention (proxy access to patient portal on bedside tablets with accompanying orientation video). A subset of parents and healthcare staff will also be interviewed about their experience with the intervention. Data will be collected through surveys, interviews, and electronic health record audits.

This study is the first multisite RCT to evaluate the impact of inpatient note access on parent-reported outcomes. By leveraging bilingual recruitment, two EHR platforms, and input from a national advisory group, the study addresses barriers to equitable access and sustainability. Findings will advance understanding of how health information technology can engage parents as partners in improving inpatient safety for children and inform broader efforts to integrate families into safety initiatives.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish-speaking parents or guardians of children under 12 years old who were hospitalized on a general pediatric service at one of the 3 centers
* Age 18 and over

Exclusion Criteria:

* Parents of children 12 years of age and older
* Parents unable to give written informed consent
* Parents of children admitted for suspected abuse or neglect
* Anticipated discharge within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of notes accessed | Duration of study participation, 2 to 7 days
  Researchers will abstract note access during hospitalization from the EHR and compare the frequency and proportion of available notes accessed between arms.

SECONDARY OUTCOMES:
Safety concern reporting | Duration of study participation, 2 to 7 days
  Safety concern reporting will be measured using the OpenNotes safety concern reporting tool, a 9-item questionnaire adapted for parent-reported safety concerns during hospitalization. The tool will be translated into Spanish and piloted for this study. Parent-reported safety concerns will be reviewed by the PI and site PIs and categorized as definite safety issues, possible safety issues, or other. Definite and possible issues will be further categorized by type (e.g., medication, physical exam) and assessed via chart reviews for associated changes to the medical record or patient care (yes/no/uncertain). Researchers will compare results across arms.
Hospital experience | Duration of study participation, 2 to 7 days
  Experience will be measured using the Child Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey, which evaluates parent perceptions of their hospital experience upon discharge. The survey includes closed-ended and Likert-style items rated on a 5-point scale, with "strongly agree" as the highest score. Key measures include overall hospital rating, willingness to recommend, and "helping you report concerns." It is available in English and Spanish. It will be administered prior to hospital discharge and compared across arms.
Change in parent activation | Baseline to discharge, 2 to 7 days
  Activation will be measured using the Parent-Patient Activation Measure (P-PAM), a 13-item Likert-style tool adapted from the Patient Activation Measure (PAM), assessing skills and confidence for managing a child's healthcare. Scores range from 0-100, with higher scores indicating greater activation. The P-PAM has demonstrated validity and reliability in both English and Spanish. It will be administered at baseline and prior to hospital discharge and compared across arms.
Change in Anxiety | Baseline to discharge, 2 to 7 days
  Anxiety will be measured using the State-Trait Anxiety Inventory (STAI) Form Y, a 40-item Likert-style questionnaire assessing anxiety on a 4-point scale. Total scores range from 20-80, with higher scores indicating greater anxiety. The STAI is validated for sensitivity to health interventions over time and is available in English and Spanish. It will be administered at baseline and prior to hospital discharge and compared across arms.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kelly, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Seattle Children's Hospital, Seattle, Washington
  - American Family Children's Hospital, Madison, Wisconsin

REFERENCES:
- [Background] O'Hare C, Gatewood AK, Baird J, Brown R, Coller RJ, Desai A, Egan A, Gerber D, McGuire T, Singh-Verdeflor KD, Smith CA, Verdelis GA, Warner G, Wong S, Kelly MM. A multicenter randomized trial to improve family clinical note access and outcomes for hospitalized children: The Bedside Notes study protocol. J Hosp Med. 2025 Nov;20(11):1256-1264. doi: 10.1002/jhm.70155. Epub 2025 Aug 21. PMID 40839550